CLINICAL TRIAL: NCT05016934
Title: Randomized Controlled-trial to Evaluate Safety, Immunogenicity and Efficacy of a Vaccine Composed of a Recombinant S1 Antigen for Prevention of Covid-19 in Adults Previously Fully Immunized With Other Vaccines
Brief Title: Evaluation of Safety and Immunogenicity of a Novel Vaccine for Prevention of Covid-19 in Adults Previously Immunized
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At collaborator's request
Sponsor: Hospital do Coracao (Other)
Collaborators: Farmacore Biotecnologia Ltda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYN 115.001.2
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A vaccine composed of a recombinant S1 antigen 10mcg (Experimental): Two applications of 10mcg of a vaccine composed of a recombinant S1 antigen 28 days apart
  Interventions: Biological: A vaccine composed of a recombinant S1 antigen
- A vaccine composed of a recombinant S1 antigen 25mcg (Experimental): Two applications of a vaccine composed of a recombinant S1 antigen 28 days apart
  Interventions: Biological: A vaccine composed of a recombinant S1 antigen
- A vaccine composed of a recombinant S1 antigen 50mcg (Experimental): Two applications of 50mcg of a vaccine composed of a recombinant S1 antigen 28 days apart
  Interventions: Biological: A vaccine composed of a recombinant S1 antigen
- Placebo (Placebo Comparator): Two applications of placebo 28 days apart
  Interventions: Biological: A vaccine composed of a recombinant S1 antigen

INTERVENTIONS:
Biological: A vaccine composed of a recombinant S1 antigen — Two applications of three different doses of a vaccine composed of a recombinant S1 antigen, a subunit of SARS-CoV-2 virus S protein

SUMMARY:
Randomized controlled trial to evaluate safety, immunogenicity and efficacy of three different doses (10, 25 and 50 mcg) of a novel vaccine compared with placebo in adult volunteers previously immunized against Covid-19 with other vaccines [Corona Vac (Sinovac), ChAdOx1 (AZ 1222, Astra Zeneca) or Ad26.Co2.S (Janssen)].

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled trial to evaluate the safety, immunogenicity and efficacy of an investigational vaccine against Covid-19 in adult volunteers previously fully immunized against Covid-19 with other vaccines [Corona Vac (Sinovac), ChAdOx1 (AZ 1222, Astra Zeneca) or Ad26.Co2.S (Janssen)].

Three different antigen doses of a vaccine composed of a recombinant S1 antigen, a subunit of SARS-CoV-2 virus S protein, will be compared against placebo to evaluate its efficacy, immunogenicity and preliminary efficacy. The study will consist of three cohorts and a total of 360 participants. Each cohort will be consisted of 120 individuals, who will be randomized in a 2:1 fashion for a vaccine composed of a recombinant S1 antigen or placebo. In the first cohort, participants will be randomized to two applications of 10mcg of a vaccine composed of a recombinant S1 antigenor placebo 28 days apart. In the first week of the study, only three volunteers will be enrolled in order to assess the safety of the vaccine after 7 days by an independent Data and Safety Monitoring Board (DSMB). The other 117 participants will be randomized only if there were no safety concerns on these three first enrolled volunteers. After the enrollment of the first 60 participants, 7-day safety data will be reviewed by the DSMB, who will decide on trial continuation sequence. If there were no safety concerns, the second cohort will start. In the second cohort, participants will be randomized to two applications of 25mcg of a vaccine composed of a recombinant S1 antigen or placebo 28 days apart. This cohort will have the same design and evaluation of safety performed on the first cohort. Again, after the enrollment of the first 60 participants, 7-day safety data will be reviewed by the DSMB, who will decide on trial continuation sequence. If there were no safety concerns, the third cohort will start. In the second cohort, participants will be randomized to two applications of 50mcg of a vaccine composed of a recombinant S1 antigen or placebo 28 days apart.

The primary endpoint of safety will be evaluated on day 7 after the first and second application of the vaccine. Therefore, all participants will have this endpoint assessed 36 days after the enrollment. The secondary endpoints will be immunogenicity, evaluated at days 29 (I.e., 28 days after the first dose) and 43 (I.e., 14 days after the second dose), and efficacy, evaluated as the incidence of symptomatic laboratory confirmed cases of Covid-19 from 14 days after the second dose until 12 months after enrollment.

A sample size was calculated based on the probability of adverse events. Assuming a 2.5% incidence of adverse events, a study with 240 participants receiving the active drug would have a probability higher than 99% to recognize at least one adverse event. Assuming a 5% incidence of adverse events, a study with 80 participants receiving the different doses (10, 25 and 50mcg) of the active drug would have a probability of 98% to recognize at least one adverse event.

As mentioned before, an independent DSMB will review safety after the enrollment of the first three participants in each cohort and again after the enrollment of the first 60 participants in each cohort. Pre-specified guidelines will be established to recommend early stopping of the trial for evidence of harm.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Previously totally immunized, I.e., two doses for Corona Vac (Sinovac) or ChAdOx1 (AZ 1222, Astra Zeneca, and one dose for Ad26.Co2.S (Janssen) vaccines at least three months before enrollment
* Negative RT-PCR for SARS-CoV-2 at the moment of triage
* No previous history of laboratory confirmed Covid-19

Exclusion Criteria:

* Pregnancy
* Participation in other vaccine trial
* Active decompensated chronic condition, namely, cardiovascular, respiratory, neurological, metabolic or hepatic diseases
* Any immunocompromise condition (primary immunodeficiencies, auto-immune diseases, long-term use of corticosteroids, solid organ transplant recipients, hematopoietic stem-cell transplant recipients, human-immunodeficiency virus active infection)
* Active cancer
* Hepatitis B or C
* History of allergic reactions to any vaccine component, including excipients and preservatives (neomycin, streptomycin, polymyxin B, eggs
* Blood donation in the past 4 weeks before screening
* Received blood product in the past 3 months before screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-04 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of local and systemic adverse events | From day 1 until day 7 after each vaccine or placebo administration
Frequency and severity of adverse events of special interest | From day 1 until day 43

SECONDARY OUTCOMES:
Quantification of interferon gamma producing T lymphocytes (INF-γ) in specific response | At days 29, 43, 91, 181 and 366
Total quantification of CD4 and CD8 T lymphocytes specific to the S1 peptide library | At days 29, 43, 91, 181 and 366
Quantification of CD4 and CD8 T lymphocytes producing specific Th1 (INF-γ, tumor necrosis factor (TNF-α) and IL-2) and Th2 (IL-4, IL-10 and IL-13) intracellular cytokines to the S1 peptide library | At days 29, 43, 91, 181 and 366
Geometric mean titer (GMT) of IgG antibody to protein S1 compared to placebo | At days 29, 43, 91, 181 and 366
Percentage of subjects with virus neutralizing antibody (NAb) in all vaccinated cases compared to placebo | At days 29, 43, 91, 181 and 366
Incidence of new cases of symptomatic laboratory confirmed by RT-PCR for SARS-CoV-2 | From day 43 to day 366

IPD SHARING:
Plan to Share IPD: No